CLINICAL TRIAL: NCT05868031
Title: Artwork in Anatomy Education: A Way to Improve Undergraduate Students' Self-efficacy and Attitude
Brief Title: Improving Undergraduate Students' Self-efficacy and Attitude by Art Work
Acronym: AAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Dr. Kevser Ozdemir, Assosiated Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SAU-FHS-KI-01
Record Dates: First submitted 2023-04-30; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Anatomy Education
Keywords: Anatomy; Education; nursing; Active learning; Artwork; Self-efficacy; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art work (Experimental): The artwork group was tasked with preparing anatomical models by hand. This hands-on approach was designed to engage the students in a more active and creative manner, allowing them to develop a deeper understanding of the subject matter. By visualizing and creating the anatomical structures themselves, the students were able to retain the information better and apply it in a practical context.
  Interventions: Other: alternative teaching methods
- Atlas groups (Experimental): The atlas group was provided with a selection of anatomical pictures from atlases and encouraged to use them as a resource to aid their learning throughout the semester. This approach focused on visual learning and aimed to provide the students with a comprehensive and detailed understanding of the anatomical structures and how they interact with one another.
  Interventions: Other: alternative teaching methods

INTERVENTIONS:
Other: alternative teaching methods — This study aimed to explore the potential benefits of alternative teaching methods in anatomy education, as well as to investigate the effectiveness of traditional lecture-based education in comparison. By examining the outcomes of these different approaches, we hope to understand better how students can best learn and retain knowledge in this field.

SUMMARY:
This study aims to evaluate the effectiveness of Artworking learning approaches in improving undergraduate students' attitudes and self-efficacy about anatomy courses.

DETAILED DESCRIPTION:
Anatomy is one of the prominent and essential disciplines in healthcare and medical education, and study the shape and structure of the body, the systems and organs that make up the body, and the relationships between these systems and organs. In health care fields, it is necessary for students to have a strong foundation in this area. However, learning anatomy can be challenging and complicated due to the complexity of the concepts and terminologies involved; it plays a crucial role in preparing future healthcare providers. (Banovac et al., 2023). Healthcare students and medical professionals need to be adequately knowledgeable about anatomy and understand the functions and spatial context of organs before performing any invasive procedures on patients (Roxburgh & Evans, 2021). Studies have shown that students without basic anatomy knowledge and skills encounter serious difficulties in advanced classes (Ghosh, 2017).

Traditional anatomy education is based predominantly on passive learning methods, such as lecture-based instruction, which may not effectively promote active student participation and knowledge retention (Ma et al., 2016). Nowadays, a revised teaching-learning approach known as active learning is implemented to ensure the curriculum remains relevant to the constantly connected and resource-rich world. It involves learners actively participating in the learning process through cooperative or hands-on tasks. Critical thinking and problem-solving skills are emphasized in this method and can improve student learning in numerous subjects (Bonatto-Costa et al., 2021). Students studying healthcare in the first year may experience challenges with the complexity and volume of anatomy subjects. However, many innovative learning tools, such as three-dimensional models, cadaver dissection, and artistic activities, such as drawing and body painting, have been conducted to enhance active learning and improve the quality of education in colleges (Rekhari & Sinnayah, 2018). Nurses and midwives rely heavily on anatomy knowledge to perform procedures such as injection sites, monitoring vital signs, administering first aid, and performing childbirth and episiotomies. A strong foundation in anatomy can facilitate professional development in these specialized areas and advanced nursing and midwifery education. Moreover, possessing a comprehensive understanding of anatomy can enhance students' self-esteem and confidence when practicing in clinical settings (Satoh et al., 2023).

Attitude refers to a student's overall evaluation of the subject, and Studies show that healthcare students have positive attitudes about anatomy during their education period. It has been believed that along with Self-efficacy, students' perspectives and attitudes toward basic science subjects, such as anatomy, can significantly affect education outcomes (Plaisant et al., 2014).

Studies show that possessing a positive attitude towards anatomy, coupled with self-efficacy, can significantly impact students' academic performance and professional development in nursing and midwifery. This underscores the importance of acquiring a strong foundation in anatomy and cultivating a positive perspective and belief in one's ability to succeed in the subject (Acar et al., 2017).

Self-efficacy is the belief in one's capability to manage and take the actions needed to succeed in learning a subject (Woolcock et al., 2016). Self-efficacy has been a leading and also reliable predictor of university student progress for years and is significantly correlated with students' grade point averages and their motivation to learn (Bartimote-Aufflick et al., 2016). Academic self-efficacy determines how well students perceive their capacity to organize and carry out courses of action related to their studies (Tembo & Ngwira, 2016).

This study aims to evaluate the effectiveness of Art working learning approaches in improving undergraduate students' attitudes and self-efficacy about anatomy courses.

Method:

This study was conducted on two groups of first-year nursing and midwifery students to compare the effectiveness of teaching anatomy using the active learning method of artwork versus anatomy atlases-based education. Questionnaires were distributed to both groups immediately after the first session of the anatomy course and 14 weeks later. The researcher responsible for distributing and collecting the questionnaires did not participate in teaching anatomy to the students. The students were asked to complete a self-report questionnaire that included information regarding their age, grade, sex, and field of study. In addition, both sets of students were also required to complete the Anatomy self-efficacy scale and Anatomy attitude scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a first-year student enrolled in Health Sciences at Sakarya University.
* Not having taken an anatomy course before.
* Being willing to participate in the research.

Exclusion Criteria:

* Not to volunteer to participate in the research.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Artwork Learning Approaches in Improving Students' Attitudes and Self-Efficacy in Anatomy Education | 14 weeks
  The outcome measure includes the assessment of anatomy self-efficacy and attitudes among the participating nursing and midwifery students. Additionally, a self-report questionnaire was administered to collect demographic information such as age, grade, sex, and field of study.
  The Anatomy Self-Efficacy Scale is a validated measurement tool that assesses students' perceived confidence in their ability to understand and apply anatomical knowledge. The Anatomy Attitude Scale is another validated measurement tool used to assess students' attitudes and beliefs toward the study of anatomy. It includes statements related to the interest, value, and enjoyment of learning anatomy.
  The data collected from the self-report questionnaire, Anatomy Self-Efficacy Scale, and Anatomy Attitude Scale will be aggregated and analyzed to evaluate the impact of different educational approaches on students' self-efficacy beliefs and attitudes towards anatomy.

CONTACTS AND LOCATIONS:
Overall Officials: kevser İlçioğlu, Dr, Principal Investigator — sakarya university, Faculty of health science, Department of nursing
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No